CLINICAL TRIAL: NCT02915354
Title: Relapse of Ankylosing Spondylitis Patients Withdrawal Etanercept After Clinical Remission: a Three Years' Following-up Study
Brief Title: Relapse of Ankylosing Spondylitis Patients Withdrawal Etanercept After Clinical Remission: a Following-up Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Gu Jieruo, Professor, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: [2006]37
Record Dates: First submitted 2016-09-23; First posted 2016-09-27 (Estimated); Last update posted 2016-11-16 (Estimated); Status verified 2016-11

CONDITIONS: Spondylitis, Ankylosing; Recurrence
MeSH Terms: conditions — Spondylitis, Ankylosing; Recurrence | interventions — Etanercept

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Etanercept, AS (Experimental): The patients were diagnosed with ankylosing spondylitis and obtained the ASAS20 response after etanercept treatment. Then they were discontinued to etanercept and received no treatment except DMARDs or NSAIDs which had used before.
  Interventions: Drug: Etanercept

INTERVENTIONS:
Drug: Etanercept — Etanercept must be discontinued. Cotherapy with disease modifying anti-rheumatic drugs or non-steroidal anti-inflammatory drugs could be continued if maintained at a stable dose for at least 4 weeks.
  Other Names: enbrel

SUMMARY:
The inclusion criteria was patients who aged 18 or older with ankylosing spondylitis, fulfilled the 1984 modified New York criteria for AS. Inclusion criteria enriched the AS patients with clinical remission, including the following definition: 1. Administration of etanercept 50 mg for 6-week period at least; 2. Acquisition of Assessment of SpondyloArthritis International Society criteria 20(ASAS20) response at the end of the treatment. We excluded patients who have developed to complete spinal fusion. We also excluded patients with kidney disease induced by other conditions; pregnancy; suckle; accompany other chronic diseases; various infections in acute stage; and other infectious diseases. At the end of the trial, patients who fulfilled the inclusions would stop etanercept treatment. Cotherapy with disease modifying anti-rheumatic drugs or non-steroidal anti-inflammatory drugs could be continued if maintained at a stable dose;Patients were followed up from the time of etanercept withdrawal per 6 weeks for 3 years by telephone. If symptoms suggestive of relapse or other problems occurred, patients were invited to come back to the center. Relapse after etanercept withdrawal was defined as an increase Bath Spondylitis Disease Activity Index(BASDAI)15 score goes back to 80 percentages of it at the beginning of the trial16. The following data were collected: demographic and disease characteristics, therapeutic modification, clinical values (BASFI, Bath Ankylosing Spondylitis Global Score (BAS-G)), Ankylosing Spondylitis Disease Activity Score (ASDAS)1718) and biologic values at baseline of the trial and the time of relapse. Adverse events and other safety measures were also collected.

DETAILED DESCRIPTION:
Patients were followed up 6 weeks by telephone. The sample size was at least 30 people. If symptoms suggestive of relapse or other problems occurred, patients were invited to come back to the center. Relapse after etanercept withdrawal was defined as an increase Bath Spondylitis Disease Activity Index(BASDAI) score goes back to 80 percentages of it at the beginning of the trial16. The following data were collected: demographic and disease characteristics, therapeutic modification, clinical values (BASFI, Bath Ankylosing Spondylitis Global Score (BAS-G)), Ankylosing Spondylitis Disease Activity Score (ASDAS) and biologic values at baseline of the trial and the time of relapse. Adverse events and other safety measures were also collected.

Demographic and baseline disease characteristics were summarized with descriptive statistics and analysed with one-way ANOVA for continuous for continuous variables and χ2 tests for categorical variables. The Kaplan-Meier method was used to estimate the time-to-relapse rate after etanercept withdrawal. Time-to-relapse curves were compared between the group of patients received 12-week and 6-week treatment of etanercept through log-rank test. The influence of the following variables including age，duration of disease, onset age, BASDAI, ASDAS-CRP, C reaction protein(CRP), and erythrocyte sedimentation rate(ESR) was examined using the Cox proportional hazards model to evaluate at etanercept withdrawal on time-to-relapse. Every continuous variable was divided into 3 categories at approximately the 33% and 67% at first19. If the relative relapse rates were not significantly different in 2 contiguous categories, they were gathered together. If no clear difference was observed in 3 categories, the median was used as a cut-off point. Normal value such as 6 mg/L for CRP level were tested. The proportional hazards model was used to study the effect of each factor on time-to-relapse and identify the independent prognostic factors. Relapse rates are presented as estimate with standard error (SE), follow-up times as median (interquartile range), and hazard ratio as estimate with 95% confidence interval.

All analyses were performed using SPSS software v16.0 (SPSS, Inc, Chicago, IL).

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of ankylosing spondylitis(1984 modified New York criteria).
* Administration of etanercept 50 mg for 6-week or 12-week.
* Acquisition of ASAS20 response at the end of the treatment.

Exclusion Criteria:

* Complete spinal fusion.
* Kidney disease induced by other conditions; pregnancy; suckle; accompany other chronic diseases; various infections in acute stage; and other infectious diseases.
* Refused to discontinue etanercept treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2007-07; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
The status of relapse | 3 years
  The cumulative probabilities of relapse at 1, 2, and 3 years were 45.7%，57.1% and 60.0%, respectively.

SECONDARY OUTCOMES:
Bath Spondylitis Disease Activity Index(BASDAI) score | 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- Rheumatology Department, the Third Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Yes
The data will be published on the Journals.

REFERENCES:
- [Background] Braun J, Sieper J. The sacroiliac joint in the spondyloarthropathies. Curr Opin Rheumatol. 1996 Jul;8(4):275-87. doi: 10.1097/00002281-199607000-00003. PMID 8864578
- [Background] de Vlam K, Mielants H, Cuvelier C, De Keyser F, Veys EM, De Vos M. Spondyloarthropathy is underestimated in inflammatory bowel disease: prevalence and HLA association. J Rheumatol. 2000 Dec;27(12):2860-5. PMID 11128677
- [Background] Braun J, de Keyser F, Brandt J, Mielants H, Sieper J, Veys E. New treatment options in spondyloarthropathies: increasing evidence for significant efficacy of anti-tumor necrosis factor therapy. Curr Opin Rheumatol. 2001 Jul;13(4):245-9. doi: 10.1097/00002281-200107000-00001. PMID 11555723
- [Background] Gorman JD, Sack KE, Davis JC Jr. Treatment of ankylosing spondylitis by inhibition of tumor necrosis factor alpha. N Engl J Med. 2002 May 2;346(18):1349-56. doi: 10.1056/NEJMoa012664. PMID 11986408
- [Background] Li ZH, Zhang Y, Wang J, Shi ZJ. Etanercept in the treatment of ankylosing spondylitis: a meta-analysis of randomized, double-blind, placebo-controlled clinical trials, and the comparison of the Caucasian and Chinese population. Eur J Orthop Surg Traumatol. 2013 Jul;23(5):497-506. doi: 10.1007/s00590-012-1035-7. Epub 2012 Jun 29. PMID 23412168
- [Background] Baji P, Pentek M, Szanto S, Geher P, Gulacsi L, Balogh O, Brodszky V. Comparative efficacy and safety of biosimilar infliximab and other biological treatments in ankylosing spondylitis: systematic literature review and meta-analysis. Eur J Health Econ. 2014 May;15 Suppl 1(Suppl 1):S45-52. doi: 10.1007/s10198-014-0593-5. Epub 2014 May 16. PMID 24832835
- [Background] Kiltz U, Baraliakos X, Braun J, van der Heijde D. Withdrawal of medical therapies in axial spondyloarthritis: what would be the optimal trial design? Clin Exp Rheumatol. 2013 Jul-Aug;31(4 Suppl 78):S47-50. Epub 2013 Oct 4. PMID 24129137
- [Background] Baraliakos X, Listing J, Brandt J, Zink A, Alten R, Burmester G, Gromnica-Ihle E, Kellner H, Schneider M, Sorensen H, Zeidler H, Rudwaleit M, Sieper J, Braun J. Clinical response to discontinuation of anti-TNF therapy in patients with ankylosing spondylitis after 3 years of continuous treatment with infliximab. Arthritis Res Ther. 2005;7(3):R439-44. doi: 10.1186/ar1693. Epub 2005 Feb 21. PMID 15899030
- [Background] Baraliakos X, Listing J, Rudwaleit M, Brandt J, Alten R, Burmester G, Gromnica-Ihle E, Haibel H, Schewe S, Schneider M, Sorensen H, Zeidler H, Visvanathan S, Sieper J, Braun J. Safety and efficacy of readministration of infliximab after longterm continuous therapy and withdrawal in patients with ankylosing spondylitis. J Rheumatol. 2007 Mar;34(3):510-5. Epub 2007 Feb 1. PMID 17299842
- [Background] Brandt J, Listing J, Haibel H, Sorensen H, Schwebig A, Rudwaleit M, Sieper J, Braun J. Long-term efficacy and safety of etanercept after readministration in patients with active ankylosing spondylitis. Rheumatology (Oxford). 2005 Mar;44(3):342-8. doi: 10.1093/rheumatology/keh475. Epub 2004 Nov 23. PMID 15561737
- [Background] Lin Q, Lin Z, Gu J, Huang F, Li T, Wei Q, Liao Z, Cao S, Jiang Y, Huang J. Abnormal high-expression of CD154 on T lymphocytes of ankylosing spondylitis patients is down-regulated by etanercept treatment. Rheumatol Int. 2010 Jan;30(3):317-23. doi: 10.1007/s00296-009-0958-8. Epub 2009 May 23. PMID 19466423
- [Derived] Zhao M, Zhang P, Fang L, Luo Z, Gu J, Lin Z. Possible predictors for relapse from etanercept discontinuation in ankylosing spondylitis patients in remission: a three years' following-up study. Clin Rheumatol. 2018 Jan;37(1):87-92. doi: 10.1007/s10067-017-3763-x. Epub 2017 Aug 7. PMID 28785857